CLINICAL TRIAL: NCT00201071
Title: Asthma Surveillance and Education in Preschool Settings
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1298; R01HL076592 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2007-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective

GROUPS / COHORTS (1):
- South Bronx, Harlem, Lower East Side

SUMMARY:
The purpose of this study is to test the effectiveness of a bilingual intervention in improving asthma care for low-income inner-city children enrolled in subsidized preschool childcare programs.

DETAILED DESCRIPTION:
BACKGROUND:

Proposed is a non-randomized, controlled, prospective trial to test the efficacy of a bilingual intervention to improve asthma care for low-income inner-city children enrolled in subsidized preschool childcare programs. Because of high rates of asthma prevalence, subsidized preschool childcare programs offer ideal settings to test innovative strategies to improve asthma care within communities at highest risk of morbidity.

DESIGN NARRATIVE:

The study will comprise three arms. Arm 1 is surveillance, in which children with asthma are identified. In Arm 2, children with asthma are identified and given written Asthma Action Plans (monitoring). Arm 3 consists of surveillance, monitoring, and education.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in specific subsidized preschools in New York City
* 2.8 to 4 years old
* Persistent asthma as defined by symptom reports
* Use of quick-relief agents or controller medications

Exclusion Criteria:

* History of intubation

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: We formed collaborative agreements with subsidized day care providers in three New York City communities with high asthma prevalence. These three communities - Harlem, the South Bronx and the Lower East Side - are economically disadvantaged communities of color. Participants were parents or guardians of children with asthma enrolled in subsidized day care center. 95% of participants were female, 64% were Hispanic, 25% were Black, 1% were White and 10% were Other. 70% were born in the continental USA, 70% spoke English as their primary language. 30% had earned less than a HS degree, 32% had received a HS diploma or a GED, 37% had attended som college, and 1% had completed college. 33% of participants had family incomes of less than $1,000 per month, 35% had incomes of $1,000 to $1,999 and 32% had incomes over $2,000.
Sampling Method: Non-Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2004-09; Primary Completion 2010-02 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Bonner, PhD, Principal Investigator — The New York Academy of Medicine, CUES
Locations (1):
- The New York Academy of Medicine, CUES, New York, New York, United States

REFERENCES:
- See also: Click here for the New York Academy of Medicine website — http://www.nyam.org